CLINICAL TRIAL: NCT04348890
Title: A Phase I/II Open-Label, Proof-of-Concept Study of Vamorolone in Children and Adolescents With Mild-Moderately Active Ulcerative Colitis
Brief Title: Proof of Concept Trial of Vamorolone in Pediatric Ulcerative Colitis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Programmatic decision
Sponsor: ReveraGen BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBP15 UC-001
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Pediatric Ulcerative Colitis
MeSH Terms: conditions — Pediatric ulcerative colitis | interventions — VBP15 compound; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: Vamorolone 4% suspension for oral dosing

INTERVENTIONS:
Drug: Vamorolone 4% suspension for oral dosing — vamorolone 6 mg/kg/day orally once daily for 8 weeks.

SUMMARY:
This is a Phase I/II, multi-center, open-label proof-of-concept study of vamorolone. Twenty participants with a flare of mild or moderately active Ulcerative Colitis (defined as a Pediatric Ulcerative Colitis Activity Index [PUCAI] 10-60) will be enrolled and receive vamorolone 6 mg/kg/day orally once daily for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent/Health Insurance Portability and Accountability Act (HIPAA) authorization prior to any study-related procedures;
* Subject has current mild to moderately active ulcerative colitis, defined as a PUCAI score of 10-60.
* Subject is ≥ 4 years old and <18 years old at the time of enrollment.
* Subject has had 1) a colonoscopy demonstrating endoscopic and histologic inflammation, and/or; 2) a fecal calprotectin > 250 mcg/g, in the preceding 1 month.
* Subject is willing and able to comply with scheduled visits, study drug administration plan, and study procedures.
* Subject has not started a new immunomodulator or biologic in the preceding 2 months.
* If subject is taking an immunomodulator and/or biologic, the dose has not been changed in the last 2 months
* Subject has a positive varicella IgG titer, or history of at least 2 documented varicella vaccines

Exclusion Criteria:

* Subject is currently being treated or has received previous treatment with oral or rectal glucocorticoids (including budesonide) in the past month
* Subject has an allergy or hypersensitivity to the study medication or to any of its constituents
* Subject has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow-up will be correctly completed or impair the assessment of study results, in the opinion of the Investigator
* Subject is taking any other investigational drug currently or has taken any other investigational drug within 3 months prior to the start of study treatment
* Clinically significant abnormal biochemical and hematological parameters, including:

  * Neutrophil count < 1000 cells/mm3
  * Platelet count ≤ 130 cells/mm3
  * Creatinine ≥ 1.2 x the upper limit of normal
  * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 2x the upper limit of normal
  * Conjugated bilirubin greater than 1.2. mg/dL
* Has active infection with enteric pathogens (including C. difficile)
* Has a positive PPD, Quantiferon Gold, or Interferon-gamma assay
* Is pregnant or breast-feeding

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Remission | 8 weeks
  Pediatric Ulcerative Colitis Activity Index score <10 and no additional therapy or colectomy). The PUCAI is scored from 0-85, lower numbers indicate less severe disease activity.

SECONDARY OUTCOMES:
Safety (adverse events) | From day 1 through 30 days after last dose
Change in osteocalcin, P1NP, CTX | From baseline to week 8 and week 12
  Bone biomarkers
Cushingoid appearance | Week 8 and Week 12
  Physician reported, yes or no
Week 8 response | Baseline to 8 Weeks and 12 Weeks
  Decrease in PUCAI score by 20 points or more (lower scores indicate less severe disease activity)
Change in Mayo Score Stool Frequency subscore | Baseline to 8 Weeks and 12 Weeks
  Score ranges from 0-3, with lower scores indicating less severe disease activity
Change in Mayo rectal bleeding score | Baseline to 8 Weeks and 12 Weeks
  Scores range from 0-3, with lower scores indicating less severe disease activity
Mayo Score Stool Frequency subscore of 0 or 1 | Week 12
Mayo Score Rectal Bleeding Score of 0 | Week 12
Change in fecal calprotectin | Baseline to Week 8 and Week 12
Change in serum C-reactive protein | Baseline to Week 8 and Week 12
Change in serum CCL22 | Baseline to Week 8 and Week 12
Change in serum miRNA 146b | Baseline to Week 8 and Week 12
Change in serum trefoil factor 3 | Baseline to Week 8 and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Conklin, MD, Study Director — ReveraGen BioPharma

IPD SHARING:
Plan to Share IPD: No